CLINICAL TRIAL: NCT07266376
Title: Validation of a VOICE MAnagement Program in Schizophrenia
Brief Title: Validation of a VOICE MAnagement Program in Schizophrenia VVoice MAPS
Acronym: PROGEVs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Collaborators: GIRCI SOHO (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PAP_RI2_2021/16
Record Dates: First submitted 2025-11-14; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Mental Disorder; Schizophrenia Diagnosis
Keywords: Schizophrenia; Auditory Verbal Hallucinations; Groupal Intervention; Integrative Approach
MeSH Terms: conditions — Mental Disorders; Schizophrenia; Hallucinations

STUDY DESIGN:
Intervention Model Description: Patients randomly assigned to the media-workshop control group will participate in 15 weekly sessions (1.5 hours each), which consist of commenting on two short episodes of the TV series Malcolm in the Middle. This early-2000s show depicts the daily life of a lower-middle-class American family. The purpose of the sessions is to enhance social cognition by practicing the reading of intentions, identifying clues supporting hypotheses, discussing these hypotheses, and considering alternative explanations.
Who Masked: Outcomes Assessor
Masking Description: Assessments will be conducted by a trained professional, blinded to the intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Media-workshop control group (No Intervention): Patients randomly assigned to the media-workshop control group will participate in 15 weekly sessions (1.5 hour per session) consisting in commenting two short episodes from the series "Malcolm in the middle". This early 2000 TV show exposes the daily life of a low middle class American family. The purpose is to focus on social cognition through the reading of intentions, identification of clues supporting any hypotheses, discuss these hypotheses or even identify alternative hypotheses.
- Psychoeducation & Metacognitive Training (Experimental): Experimental group sessions are organized as follow : Psychoeducation of AVHs (sessions 1 and 2); Metacognitive training (sessions 3 to 6); Paying attention to voices through the use of a notebook (sessions 7 to 9); Taking control over the voices through - Attentional Distraction (session 10); Voice avatar creation (session 11); Dialogue with voices (sessions 12 & 13); Compassion-based mindfulness (session 14); Living with voices and community integration (session 15).
  Interventions: Behavioral: Integrative group therapy

INTERVENTIONS:
Behavioral: Integrative group therapy — Integrative group therapy includes 15 sessions weekly, 1.5 hours sessions supervised by one psychologist and one nurse, trained in or at least familiar with cognitive-behavioural therapy.
  Arms: Psychoeducation & Metacognitive Training

SUMMARY:
Approximately 25-50% of patients with schizophrenia experience treatment-resistant Auditory Verbal Hallucinations (AVHs), which contribute to the development of associated psychopathological disorders (e.g., anxiety, depression, suicidal ideation). Various validated psychotherapeutic strategies and tools for managing treatment-resistant AVHs have been combined into an integrative therapeutic program. The main objective of this study is to evaluate the efficacy of this program in reducing the frequency and intensity of AVHs, as well as its impact on comorbid psychopathology (e.g., depression, anxiety, self-esteem, substance use) in patients with schizophrenia or schizoaffective disorder who experience treatment-resistant AVHs.

DETAILED DESCRIPTION:
The present study is a multicenter, prospective, randomized trial with two groups. Its main objective is to evaluate the efficacy of an integrative group therapy for drug-resistant Auditory Verbal Hallucinations (AVHs) in patients with schizophrenia or schizoaffective disorder. A total of 114 patients will be randomly assigned to the experimental or control group. The experimental group will receive integrative therapy sessions, while the control group will participate in an audio-visual group reflecting usual care.

Both experimental and control groups will attend fifteen weekly 1.5-hour sessions, supervised by a psychologist and a nurse trained in, or at least familiar with, cognitive-behavioral therapy. The sessions for the experimental group are organized as follows:

Sessions 1-2: Psychoeducation about AVHs Sessions 3-6: Metacognitive training Sessions 7-9: Monitoring voices using a notebook Session 10: Gaining control over voices through attentional distraction Session 11: Voice avatar creation Sessions 12-13: Dialogue with voices Session 14: Compassion-based mindfulness Session 15: Living with voices and community integration

ELIGIBILITY:
Inclusion Criteria

Consenting patients over 18 years of age will be enrolled in the study if they meet all of the following criteria:

* Diagnosis: Fulfill DSM-5 criteria for schizophrenia or schizoaffective disorder.
* Resistant AVHs: Present treatment-resistant auditory verbal hallucinations (AVHs), defined as the persistence of daily hallucinations without remission despite adequate antipsychotic medication for at least 3 months.
* Motivation: Express a request for relief from voices.
* Treatment Setting: Are outpatients being treated in psychiatric departments at the Public Mental Health Institution of Guadeloupe or the University Hospital Center of Nîmes.
* Severity: Have a score of greater than 9 on the Psychotic Symptom Rating Scale - Auditory Hallucinations subscale (PSYRATS-AH).

Exclusion Criteria :

Patients will be excluded from the study if they meet any of the following criteria:

* Participation in another study: Currently taking part in another clinical trial or within the exclusion period of another study.
* Consent refusal: Refuse to sign the written informed consent.
* Inability to provide informed consent: Failure or impossibility to provide the patient with sufficient information to allow an informed decision.
* Severe substance abuse: Presence of severe substance use disorder.
* Acute somatic decompensation: Experiencing an acute medical condition that may compromise participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2027-01-05 (Estimated); Study Completion 2027-01-05 (Estimated)

PRIMARY OUTCOMES:
Change in Phenomenological Features of Auditory Verbal Hallucinations (AVHs) | Baseline (before the intervention, D1), one month after the end of the intervention (D2), and six months after the end of the intervention (D3).
  Change in Phenomenological Features of Auditory Verbal Hallucinations (AVHs) Changes in the severity, intensity, frequency, and associated distress of AVHs will be assessed using the Psychotic Symptom Rating Scale - Auditory Hallucinations subscale (PSYRATS-AH).
  The PSYRATS-AH includes 11 items, each rated on a 0-4 Likert scale (total score range: 0 to 44), where higher scores indicate more severe hallucination-related symptomatology.
  All evaluations will be performed by an investigator blinded to group allocation to ensure unbiased assessment of treatment effects.

SECONDARY OUTCOMES:
Belief and Trust in AVHs | Baseline (D1), one month after the end of the intervention (D2), and six months after the end of the intervention (D3).
  Belief and Trust in Auditory Verbal Hallucinations (AVHs) Beliefs about and trust in AVHs will be assessed using the Beliefs About Voices Questionnaire-Revised (BAVQ-R). The BAVQ-R evaluates participants' beliefs, emotional responses, and behavioral engagement with voices. Each item is rated on a 0-4 Likert scale, with a total score range of 0 to 56, where higher scores indicate stronger beliefs in, or greater trust toward, the voices.
  All assessments will be conducted by an investigator blinded to group assignment to ensure unbiased evaluation.
Attitudes and Reactions Towards AVHs | Baseline (D1), one month after the end of the intervention (D2), and six months after the end of the intervention (D3).
  Attitudes and Reactions Towards Auditory Verbal Hallucinations (AVHs) Attitudes toward and behavioral reactions to AVHs will be assessed using the Voice Attitude and Action Scale - 9 items (VAAS-9). Each item is rated on a 0-4 Likert scale, resulting in a total score range of 0 to 36, where higher scores indicate more adaptive attitudes and actions toward voices.
  All assessments will be performed by an investigator blinded to group assignment to ensure unbiased measurement.
Depression | Baseline (D1), one month after the end of the intervention (D2), and six months after the end of the intervention (D3).
  Depressive symptoms will be assessed using the Calgary Depression Scale for Schizophrenia (CDSS). The CDSS consists of 9 items, each scored on a 0-3 scale, resulting in a total score range of 0 to 27, where higher scores indicate more severe depressive symptoms.
  All assessments will be conducted by an investigator blinded to group assignment to ensure unbiased evaluation.
Self-Esteem | Baseline (D1), one month after the end of the intervention (D2), and six months after the end of the intervention (D3).
  Self-esteem will be assessed using the Rosenberg Self-Esteem Scale (RSES). The scale includes 10 items, each rated on a 0-3 Likert scale, resulting in a total score range of 0 to 30, where higher scores indicate higher self-esteem.
  All assessments will be conducted by an investigator blinded to group assignment to ensure unbiased measurement.
Subjective Quality of Life | Baseline (D1), one month after the end of the intervention (D2), and six months after the end of the intervention (D3).
  Subjective quality of life will be assessed using the World Health Organization Quality of Life Instrument - WHOQOL-BREF. The WHOQOL-BREF includes 26 items across four domains (physical health, psychological health, social relationships, and environment), with each item rated on a 1-5 Likert scale, resulting in domain scores that can be transformed to a 0-100 scale, where higher scores indicate better quality of life.
  All assessments will be conducted by an investigator blinded to group assignment to ensure unbiased evaluation.
Exploratory Outcome: Substance Use | Baseline (D1 - before intervention); One month after the end of the intervention (D2); Six months after the end of the intervention (D3)
  Changes over time in substance use will be assessed using the Alcohol, Smoking and Substance Involvement Screening Test - Version 3 (ASSIST V3.0). The ASSIST V3.0 evaluates the frequency and risk level of substance use across multiple substances (e.g., alcohol, tobacco, cannabis, cocaine, opioids, stimulants, sedatives). Each item is scored according to substance-specific guidelines, resulting in risk scores ranging from 0 to 39 for each substance, where higher scores indicate greater risk or more severe substance use involvement.
  All assessments will be conducted by an investigator blinded to group assignment to ensure unbiased evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Jumentier, PhD, Study Director — Public Mental Health Institution of Guadeloupe
Locations (1):
- Public Mental Health Institution of Guadeloupe, Les Abymes, Guadeloupe